CLINICAL TRIAL: NCT04315376
Title: Exercise Program and Diet Intervention Attenuated Inflammation Through Down-regulation of ASC Gene and Inflammatory Markers in Obese Adults
Brief Title: Exercise and Diet Intervention Attenuated Inflammation Through ASC Gene and Inflammatory Markers in Obese Adults
Acronym: INDIEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, ERIKA MARTINEZ-LOPEZ, Study director, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI-08518
Record Dates: First submitted 2020-03-15; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Inflammatory Response; Obesity; Abdominal Obesity; Diet Habit; Exercise
Keywords: Nutrition; Exercise; Diet; Inflammation; Obesity
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Feeding Behavior; Motor Activity; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise-Diet Group (Experimental): The participants receive a personal exercise program according to Astrand-rhyming test baseline results, and a hypo-caloric diet intervention
  Interventions: Behavioral: Exercise-Diet Intervention
- Diet Group (Active Comparator): The participants no receive a personal exercise program, only the hypo-caloric diet
  Interventions: Behavioral: Diet Intervention

INTERVENTIONS:
Behavioral: Exercise-Diet Intervention — The participants who performed exercise-diet intervention performed an Astrand-rhyming test before and after the exercise program intervention. Participants followed a progressive exercise-program during four months according to initial physical fitness. The main exercises consisted of improving aerobic, speed and resistance performance. During all single sessions, breathlessness and fatigue were measured using 0 to10 Borg scale. A personal trainer certified by American College of Sports Medicine (ACSM) supervised three sessions per week, the other two unsupervised training days the subjects were given the detailed training program to do in house/park. And also, this group received a diet intervention that consisted of a 20 percentage reduction of total energy expenditure estimated by the Mifflin formula with a nutrients distribution as follows: 50% carbohydrates, 30% lipids, and 20% proteins.
  Arms: Exercise-Diet Group
Behavioral: Diet Intervention — This group received a diet intervention that consisted of a 20 percentage reduction of total energy expenditure estimated by the Mifflin formula with a nutrients distribution as follows: 50% carbohydrates, 30% lipids, and 20% proteins.
  Arms: Diet Group

SUMMARY:
Background: Obesity is one of the most important health problems worldwide, several factors related to lifestyle as physical inactivity and unbalanced diets increase their development. This condition is characterized by low-chronic inflammation by excess of adipose tissue. The apoptosis-associated speck-like protein containing a caspase recruitment domain (ASC) protein is part of NLRP3 inflammasome, a complex related to inflammation and metabolic alterations.

Purpose: The aim of this study was to evaluate the effect of physical exercise program on ASC gene expression and inflammatory markers in obese adults.

Methods: 37 obese individuals were randomized to exercise-diet group or diet-group during a 4-month follow-up period. The dietary evaluation was analyzed by Nutritionist Pro software. Body composition was evaluated by bioimpedance (InBody 370). All biochemical determinations were analyzed by dry chemistry (Vitros 350). ASC messenger ribonucleic acid (mRNA) expression was performed by real-time polymerase chain reaction (PCR) using Taqman probes and by the 2-ΔΔcq quantification method. Cytokine levels was performed using the Bio-PlexPro™ HumanTh17Cytokine Assays (MagPix) panel. Statistical analysis was performed with Statistical Package for the Social Sciences (SPSS) v.22 software.

DETAILED DESCRIPTION:
A randomized clinical trial was conducted in the Institute of Translational Nutrigenetics and Nutrigenomics, Department of Molecular Biology in Medicine, Health Sciences Center, at the University of Guadalajara, Guadalajara, Jalisco, Mexico, from February of 2018 to February of 2019. All participants were recruited through flyers and social media invitations. Sample size was determined according to the mean difference formula for clinical trials. To achieve a statistical power of 80% and an alpha of 5%, a sample size of 13 participants in each study group was required. However, 37 obese individuals who met the selection criteria were randomized in exercise-diet group or diet-group. Blood sample, height and weight were measured after 8-12 hour fast and wearing light clothes. The participants in the exercise-diet group were cited in the Respiratory Unit of the University of Guadalajara with the indication of not consuming caffeine, tobacco or energy drinks 24 hours before the test, and not having eaten food at least two hours before the Astrand-rhyming Test. This study was approved by the Ethics and Biosafety Committee of the Health Sciences Center, University of Guadalajara (registry number CUCS/CINV/0476/18). The procedures were in accordance with this institution's guidelines and all the participants signed a written consent-informed.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than 30 kg/m^2
* Sedentary individuals
* Both genres
* Waist circumference greater than 80 centimeters in women and greater than 90 centimeters in men

Exclusion Criteria:

* Pregnant or breastfeeding women
* Diagnosis of any metabolic disease or cancer
* Alcohol or tobacco consumption
* Muscle or joint injury

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Change in ASC mRNA Expression | Mean change from baseline (0 Month) to end of treatment at 4th Month.
  The polymorphonuclear cells were separated using Dextran treatment from peripheral blood samples. Subsequently, TRIzol® reagent was using according to the manufacturer´s instructions. The complementary DNA (cDNA) synthesis was performed according to standard techniques.
  Quantitative real-time PCR was performed using TaqMan® probes in Light Cycler 96 equipment considering standards PCR conditions to analyze ASC mRNA relative expression by 2-ΔΔcq method. The amplification reactions were performed in duplicate using β-Actin gene as constitutive gene to normalized the samples.
Change in Pro-inflammatory and Anti-inflammatory Cytokines | Mean change from baseline (0 Month) to end of treatment at 4th Month.
  The pro-inflammatory and anti-inflammatory cytokines quantification were using Bio-Plex Pro™ Human cytokine Standard 17-Plex, Group I kit following the supplier's instructions, and the read was immediately by MAGPIX™ analyzer.
Change in Astrand-rhyming Submaximal Test | Mean change from baseline (0 Month) to end of treatment at 4th Month.
  The Astrand-rhyming submaximal test was performed as described by Astrand.

SECONDARY OUTCOMES:
Changes in Height | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month. 1st month, 2nd month, 3th month and the 4th month.
  Height in meters using a stadiometer.
Changes in Weight | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month.
  The weight was measured in kilograms on InBody 370.
Changes in Body Mass Index (BMI) | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month.
  Weight and height were be combined to report BMI in kg/m^2
Changes in Waist Circumference | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month.
  Waist circumference was measured at the narrowest point between the edge of the inner rib and the iliac crest, with the participant in an abducted and relaxed position, after expiration using a Lufkin Executive® tape.
Changes in Fat Mass | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month.
  The Fat Mass was measured in kilograms by electrical bioimpedance on InBody 370.
Changes in Musculoskeletal Mass | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month.
  The musculoskeletal mass was measured in kilograms by electrical bioimpedance on InBody 370.
Changes in Serum Glucose | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month.
  It was measured in mg/dL using a dry chemistry system in Vitros 350 equipment.
Changes in Serum Insulin | At the baseline (0 Month), 3th month and the 4th month.
  Were determined through Insulin Model ELISA kit following the supplier's instructions.
Changes in homeostatic model assessment - insulin resistance (HOMA-IR) | At the baseline (0 Month), 3th month and the 4th month.
  Serum glucose and Insulin levels were be combined to report HOMA-IR calculated as described by Matthews.
Changes in Total Cholesterol | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month.
  It was measured in mg/dL using a dry chemistry system in Vitros 350 equipment.
Changes in High-density lipoprotein (c-HDL) | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month.
  It was measured in mg/dL using a dry chemistry system in Vitros 350 equipment.
Changes in Atherogenic Index | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month.
  Serum total cholesterol and c-HDL were be combined to report atherogenic index, calculated through formula [Total cholesterol (mg/dL) / HDL-c (mg/dL)].

CONTACTS AND LOCATIONS:
Overall Officials: Erika Martínez-López, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Erika Martínez-López, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared to protect and safeguard the confidentiality data of the participants.

REFERENCES:
- [Result] ASTRAND PO, RYHMING I. A nomogram for calculation of aerobic capacity (physical fitness) from pulse rate during sub-maximal work. J Appl Physiol. 1954 Sep;7(2):218-21. doi: 10.1152/jappl.1954.7.2.218. No abstract available. PMID 13211501
- [Result] Lin CH, Chiang SL, Tzeng WC, Chiang LC. Systematic review of impact of lifestyle-modification programs on metabolic risks and patient-reported outcomes in adults with metabolic syndrome. Worldviews Evid Based Nurs. 2014 Dec;11(6):361-8. doi: 10.1111/wvn.12069. PMID 25488565
- [Result] Ozaki E, Campbell M, Doyle SL. Targeting the NLRP3 inflammasome in chronic inflammatory diseases: current perspectives. J Inflamm Res. 2015 Jan 16;8:15-27. doi: 10.2147/JIR.S51250. eCollection 2015. PMID 25653548
- [Result] Ross R, Hudson R, Stotz PJ, Lam M. Effects of exercise amount and intensity on abdominal obesity and glucose tolerance in obese adults: a randomized trial. Ann Intern Med. 2015 Mar 3;162(5):325-34. doi: 10.7326/M14-1189. PMID 25732273
- [Result] Taniguchi S, Sagara J. Regulatory molecules involved in inflammasome formation with special reference to a key mediator protein, ASC. Semin Immunopathol. 2007 Sep;29(3):231-8. doi: 10.1007/s00281-007-0082-3. Epub 2007 Sep 6. PMID 17805543
- [Result] You T, Arsenis NC, Disanzo BL, Lamonte MJ. Effects of exercise training on chronic inflammation in obesity : current evidence and potential mechanisms. Sports Med. 2013 Apr;43(4):243-56. doi: 10.1007/s40279-013-0023-3. PMID 23494259
- [Derived] Barron-Cabrera E, Gonzalez-Becerra K, Rosales-Chavez G, Mora-Jimenez A, Hernandez-Canaveral I, Martinez-Lopez E. Low-grade chronic inflammation is attenuated by exercise training in obese adults through down-regulation of ASC gene in peripheral blood: a pilot study. Genes Nutr. 2020 Aug 27;15(1):15. doi: 10.1186/s12263-020-00674-0. PMID 32854610